CLINICAL TRIAL: NCT01371357
Title: The Effects of 8-week Choline, Betaine, and Folic Acid Supplementation on Plasma Homocysteine Concentration During Guanidinoacetic Acid Loading in Young Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Sergej M. Ostojic, MD, PhD, Head of Exercise Physiology Lab, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN-214E-S10
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Hyperhomocysteinemia
Keywords: Remethylation; Human Subjects; Clinical Trial; B-vitamin; Creatine
MeSH Terms: conditions — Hyperhomocysteinemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TEST1 (Experimental): 2.4 g/day of guanidinoacetic acid
  Interventions: Drug: TEST 1
- TEST 2 (Experimental): 2.4 g/day of guanidinoacetic acid + 3.0 g/day of choline dihydrogen citrate + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Interventions: Drug: TEST 2
- TEST 3 (Experimental): 2.4 g/day of guanidinoacetic acid + 1.6 g/day of betaine HCl + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Interventions: Drug: TEST 3
- TEST 4 (Experimental): 2.4 g/day of guanidinoacetic acid + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Interventions: Drug: TEST 4

INTERVENTIONS:
Drug: TEST 1 — 2.4 g/day of guanidinoacetic acid
  Arms: TEST1
Drug: TEST 2 — 2.4 g/day of guanidinoacetic acid + 3.0 g/day of choline dihydrogencitrate + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Arms: TEST 2
Drug: TEST 3 — 2.4 g/day of guanidinoacetic acid + 1.6 g/day of betaine HCl + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Arms: TEST 3
Drug: TEST 4 — 2.4 g/day of guanidinoacetic acid + 5 µg/day of B12 + 10 mg/day of B6 + 600 µg/day of folic acid
  Arms: TEST 4

SUMMARY:
A methyl-group acceptor such as guanidinoacetic acid (GAA) could induce hyperhomocysteinemia with the effects of GAA expected to be dose-dependent. Due to the fact that hyperhomocysteinemia is thought to be an independent risk factor for cardiovascular and neurodegenerative diseases, different dietary agents were used in the past for the treatment of elevated total plasma homocysteine (T-HCy), e. g. betaine, choline (betaine precursor) or folic acid. In the context of GAA loading the question arises whether intake of betaine, choline (betaine precursor) or folic acid during GAA loading could affect plasma T-HCy in healthy humans. Forty healthy physically active men and women aged 20 to 30 years will take part in this GAA-controlled, double-blind and parallel-group intervention study. Subjects will be allocated to four randomly assigned trials, with treatment lasting for 8 weeks and washout period of 28 days. The 4 test treatment-groups will include TEST1 (GAA only), TEST2 (GAA, choline, B6, B12 and folic acid), TEST3 (GAA, betaine, B6, B12 and folic acid) and TEST4 (GAA, B6, B12 and folic acid). Plasma T-HCy will be the primary outcome measure assessed every second week throughout the study. Plasma B-vitamins and blood and urine metabolites (GAA, creatine, methionine, arginine) will be secondary outcome measures along with adverse-effects indicators assessed every second week throughout the study. Selected body composition indicators will be obtained at 0, 2, 8 and 12 weeks throughout the study to monitor the effects of experimental treatments on body hydration and protein synthesis. This research will test the hypothesis that a combination of GAA with homocysteine lowering nutrients attenuates the elevation of T-hcy, and will further display the size-effect of each additive used.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and non-pregnant females
* moderately physically active
* aged 20 to 30 years
* not currently taking any dietary supplement for the past 2 months

Exclusion Criteria:

- total plasma homocysteine above 15.5 µmol/L

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Total plasma homocysteine | 3 months

SECONDARY OUTCOMES:
Serum creatine | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Center for Health, Exercise and Sport Sciences
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia

REFERENCES:
- [Background] Olthof MR, Brink EJ, Katan MB, Verhoef P. Choline supplemented as phosphatidylcholine decreases fasting and postmethionine-loading plasma homocysteine concentrations in healthy men. Am J Clin Nutr. 2005 Jul;82(1):111-7. doi: 10.1093/ajcn.82.1.111. PMID 16002808
- [Background] Setoue M, Ohuchi S, Morita T, Sugiyama K. Hyperhomocysteinemia induced by guanidinoacetic acid is effectively suppressed by choline and betaine in rats. Biosci Biotechnol Biochem. 2008 Jul;72(7):1696-703. doi: 10.1271/bbb.70791. Epub 2008 Jul 7. PMID 18603787
- [Background] Verhoef P, de Groot LC. Dietary determinants of plasma homocysteine concentrations. Semin Vasc Med. 2005 May;5(2):110-23. doi: 10.1055/s-2005-872397. PMID 16047264